CLINICAL TRIAL: NCT02471352
Title: Studies of Dermatologic Diseases-Biospecimen Acquisition Protocol
Brief Title: Studies of Dermatologic Diseases Biospecimen Acquisition Protocol
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150144; 15-AR-0144
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Dermatologic Conditions; Healthy Volunteers; Normal Volunteers; Carcinoma, Merkel Cell
Keywords: Dermatologic Condition; Skin Disease; Biospecimen; Healthy Volunteers; Merkel Cell Carcinoma; Natural History
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/ Skin disease or at risk: Subjects with a skin disease or at risk of developing a skin disease/ Family member of persons with a skin disease
- 2/ Healthy Volunteers: Healthy Volunteers

SUMMARY:
Background:

- Skin disease can have many causes. It can have widespread consequences, and in rare cases can lead to death. Researchers want to determine the causes of various types of skin diseases and find a way to treat them.

Objectives:

- To determine the causes of various skin diseases and find ways to treat them.

Eligibility:

* People ages 2 and older who have:

  * A skin disease or at risk of developing a skin disease OR
  * A family member of persons with a skin disease
* Healthy volunteers ages 2 and older

Design:

* Participants will be screened under a separate protocol.
* Participants may take a survey about how their skin condition affects their quality of life.
* Participants will have a medical history and a physical exam including a detailed skin exam. Pictures will be taken of their skin to document any skin disease.
* Participants will have specimens collected. This may include:

  * Several teaspoons of blood taken at each visit
  * Stool samples
  * Nail and body fluid (like saliva) samples
  * Cheek swabs. The inside of the cheek will be scraped for about a minute in each direction to collect cells.
  * Collection of skin samples with:

    * A swab (like a Q-tip)
    * Gently scraping skin to remove the outer layers of cells
    * Applying and removing 1-inch pieces of tape
* Participants may have up to 4 skin biopsies in 12 months, with 4 separate biopsies taken each time.

  * An area of skin will be numbed with an injection.
  * A piece of skin the size of a pencil eraser will be removed using a small instrument.
  * A flat scar usually develops at the biopsy site.

DETAILED DESCRIPTION:
Background:

* Skin diseases represent one of the most common medical problems in the United States, affecting 1 in 3 people at any given time.
* Complex interactions between genetic background and the environment are relevant to understanding skin disease.
* By studying dermatoses, we may gain insight into the complex host-environment interactions that give rise to or exacerbate these skin conditions, and into links between inflammation and cancer.

Objective:

-To procure biologic samples for exploratory cellular, molecular, genetic and genomic biological studies from subjects with dermatologic conditions, subjects at risk for developing dermatologic conditions and healthy volunteers in the support of NIH biomedical studies

Eligibility:

-Subjects with or at risk for developing dermatologic diseases, family members of subjects with dermatologic diseases, or healthy volunteers, including adults and children.

Design:

* The purpose of this study is to examine, in an exploratory fashion, a variety of biologic assays relevant to the investigation of dermatologic diseases.
* Approximately 50 subjects are anticipated to consent to the study each year with an accrual ceiling of 700 consented subjects planned over 10 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Eligible participants must:

  * Have a dermatologic condition, as determined by the PI or AIs, OR --be at risk for developing a dermatologic condition, as determined by the PI or AIs, OR
  * be a family member of a person with a dermatologic condition OR
  * be a healthy volunteer, as defined as a person with no known significant health problems.
  * Be willing to provide biospecimens for research and clinical studies, and for storage to be used for future research.
  * Subjects of age greater than 0 years old (including only viable neonates) are eligible.

EXCLUSION CRITERIA:

* Presence of conditions that, in the judgment of the investigator, may put the subject at undue risk or make them unsuitable for participation in the study.
* Inability to comply with the requirements of the protocol.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Referrals of eligible subjects currently undergoing evaluation and/or treatment at the NIH Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-06-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Procure biologic samples for exploratory cellular, molecular, genetic and genomic biological studies | Time of collection
  Collection of biologic samples

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on sharing IPD.

REFERENCES:
- [Derived] Ahmed N, Joglekar P, Deming C; NISC Comparative Sequencing Program; Lemon KP, Kong HH, Segre JA, Conlan S. Genomic characterization of the C. tuberculostearicum species complex, a prominent member of the human skin microbiome. mSystems. 2023 Dec 21;8(6):e0063223. doi: 10.1128/msystems.00632-23. Epub 2023 Nov 10. PMID 38126779
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-AR-0144.html